CLINICAL TRIAL: NCT01926808
Title: Vitamin D Serum Concentrations and Vitamin D Supplementation in Children and Young Adults With Cerebral Palsy
Brief Title: Vitamin D Serum Concentrations & Supplementation in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Martha Blackford, PharmD, PharmD, Akron Children's Hospital
Other Study IDs: Longitudinal Vitamin D
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitamin D supplementation

SUMMARY:
The purpose of this study is to try to correlate vitamin D dosing and dosing adjustment with Vitamin D levels, measure affects of seizure medications on levels as well as pathologic fractures and bone density in severely cognitively impaired, non-mobile children and adolescents with CP.

ELIGIBILITY:
Inclusion Criteria:

* Recorded vitamin D supplementation dose (i.e. prescribed diet and any additional sources of vitamin D) with at least two serum vitamin D concentrations recorded in the medical chart from January 1, 2008 to June 30, 2013.
* Resident of HLCCD since 2008

Exclusion Criteria:

* No vitamin D levels recorded.
* History of hyperthyroidism or parathyroid pathology.
* Short gut syndrome that requires TPN.
* Poor medical documentation.
* Heritable disorders that affect vitamin D levels such as Pseudovitamin D deficiency rickets, Vitamin D resistant rickets, autosomal dominant hypophosphatemic rickets and X-linked hypophosphatemic rickets

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Severely cognitively impaired, non-mobile children and young adults who are residents at long-term care facility
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in serum vitamin D concentrations | 5 years